CLINICAL TRIAL: NCT00534235
Title: Post-Approval Study to Investigate The Long Term (5-Year) Survivorship of Coflex Compared to Control Fusion Study Patients
Brief Title: Post-Approval Clinical Trial Comparing the Long Term Safety and Effectiveness Coflex vs. Fusion to Treat Lumbar Spinal Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paradigm Spine (Industry)
Collaborators: MCRA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PS-001
Record Dates: First submitted 2007-09-20; First posted 2007-09-24 (Estimated); Results first posted 2019-02-27 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-01

CONDITIONS: Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis | interventions — Decompression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Posterolateral Fusion w/Pedicle Screws (Active Comparator): Control: Posterolateral fusion and implantation of pedicle screws after decompression
  Interventions: Procedure: Decompression; Device: Posterolateral Fusion and Implantation of Pedicle Screws
- coflex Interlaminar Technolgy (Active Comparator): Investigative: Implantation of coflex Interlaminar Technology after decompression
  Interventions: Procedure: Decompression; Device: Implantation of coflex Interlaminar Technology

INTERVENTIONS:
Procedure: Decompression — Either microsurgical decompression or laminotomy to remove bone impinging on nerves causes the patient pain
Device: Posterolateral Fusion and Implantation of Pedicle Screws
  Arms: Posterolateral Fusion w/Pedicle Screws
Device: Implantation of coflex Interlaminar Technology
  Arms: coflex Interlaminar Technolgy

SUMMARY:
Post-Approval Clinical Study Comparing the Long Term Safety and Effectiveness of coflex vs. Fusion to Treat Lumbar Spinal Stenosis

DETAILED DESCRIPTION:
The primary objective of this post-approval study is to examine the long-term survivorship of the coflex®. The coflex® Interlaminar Technology is an interlaminar stabilization device indicated for use in one or two level lumbar stenosis from L1-L5 in skeletally mature patients with at least moderate impairment in function, who experience relief in flexion from their symptoms of leg/buttocks/groin pain, with or without back pain, and who have undergone at least 6 months of non-operative treatment. The coflex® is intended to be implanted midline between adjacent lamina of 1 or 2 contiguous lumbar motion segments. Interlaminar stabilization is performed after decompression of stenosis at the affected level(s).

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2012-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Davis R, Auerbach JD, Bae H, Errico TJ. Can low-grade spondylolisthesis be effectively treated by either coflex interlaminar stabilization or laminectomy and posterior spinal fusion? Two-year clinical and radiographic results from the randomized, prospective, multicenter US investigational device exemption trial: clinical article. J Neurosurg Spine. 2013 Aug;19(2):174-84. doi: 10.3171/2013.4.SPINE12636. Epub 2013 May 31. PMID 23725394
- See also: Related Info — http://www.paradigmspine.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Posterolateral Fusion w/Pedicle Screws: Control: Posterolateral fusion and implantation of pedicle screws after decompression
  Decompression: Either microsurgical decompression or laminotomy to remove bone impinging on nerves causes the patient pain
  Posterolateral Fusion and Implantation of Pedicle Screws
- Coflex Interlaminar Technolgy: Investigative: Implantation of coflex Interlaminar Technology after decompression
  Decompression: Either microsurgical decompression or laminotomy to remove bone impinging on nerves causes the patient pain
  Implantation of coflex Interlaminar Technology
Period: Overall Study
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Started | 107 | 215
Completed | 91 | 192
Not Completed | 16 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy | Total
Number analyzed (Participants) | 107 | 215 | 322
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (9.0) | 62.1 (9.2) | 62.8 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 106 | 164
  Male | 49 | 109 | 158
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian / Alaskan Native | 3 | 1 | 4
  Asian | 3 | 4 | 7
  Black or African American | 6 | 11 | 17
  White | 93 | 191 | 284
  Other | 2 | 8 | 10
Region of Enrollment [Number; unit: participants]
  United States | 107 | 215 | 322
Weight [Mean (Standard Deviation); unit: pounds] | 187.7 (38.1) | 190.3 (35.4) | 189.5 (36.3)
Height [Mean (Standard Deviation); unit: inches] | 66.6 (4.1) | 67.0 (4.1) | 66.9 (4.1)
Current Smoker [Count of Participants; unit: Participants]
  Yes | 15 | 22 | 37
  No | 92 | 193 | 285
Comorbidities [Count of Participants; unit: Participants]
  Cardiovascular | 74 | 137 | 211
  Musculoskeletal | 61 | 112 | 173
  Endocrine | 35 | 55 | 90
Duration of Back Pain [Count of Participants; unit: Participants]
  None | 0 | 0 | 0
  Fewer than 6 months | 1 | 3 | 4
  6 months to a year | 14 | 24 | 38
  More than one year | 92 | 188 | 280
Duration of Leg Pain (maximum) [Count of Participants; unit: Participants]
  None | 1 | 1 | 2
  Fewer than 6 months | 8 | 6 | 14
  6 months to a year | 22 | 38 | 60
  More than one year | 76 | 170 | 246
Duration of Buttock Pain [Count of Participants; unit: Participants]
  None | 21 | 32 | 53
  Fewer than 6 months | 7 | 11 | 18
  6 months to a year | 22 | 41 | 63
  More than one year | 57 | 131 | 188
Duration of Groin Pain [Count of Participants; unit: Participants]
  None | 74 | 157 | 231
  Fewer than 6 months | 5 | 6 | 11
  6 months to a year | 12 | 13 | 25
  More than one year | 16 | 39 | 55

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Improvement of at Least 15 Points in ODI
Description: The primary variable of performance is the assessment of Oswestry Low Back Pain Disability Index (ODI) in both treatment groups at 5 years. It will be assessed if the improvement in ODI since the pre surgery status in the coflex™ group is better than the improvement in the control group (scale 0-100 with a higher score representing increased disability).
Time Frame: 5 years
Population: The accounting #s in the Patient Flow include all subjects available for CCS evaluation; therefore, the overall # of participants analyzed for each Outcome Measure will differ from the number provided in the Participant Flow as the number provided for each Outcome Measure is the number of patients who completed or were assessed for that measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 54 | 126
Participants | 41 | 101

2. Primary Outcome: Number of Subjects With no Reoperations, Revisions, Removals, or Supplemental Fixation
Description: Assessment of secondary surgical interventions, i.e., reoperations, revisions, removals, or supplemental fixation associated with either coflex or control group. Refer to FDA guidance for complete definitions (https://www.fda.gov/RegulatoryInformation/Guidances/ucm072263.htm).
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 107 | 215
Participants | 87 | 179

3. Primary Outcome: Number of Subjects With no Major Device Related Complications
Description: Assessment of major device-related complications at 5 years
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 107 | 215
Participants | 100 | 212

4. Primary Outcome: Number of Subjects With no Epidural Injection(s)
Description: Assessment of lumbar epidural injections
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 107 | 215
Participants | 84 | 177

5. Primary Outcome: Number of Subjects With no Persistent New or Increasing Sensory or Motor Deficit
Description: No persistent new or increasing sensory or motor deficit
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 74 | 145
Participants | 70 | 135

6. Primary Outcome: Number of Subjects With no Persistent New or Increasing Sensory Deficit
Description: No persistent new or increasing sensory deficit
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 75 | 146
Participants | 72 | 137

7. Primary Outcome: Number of Subjects With no Persistent New or Increasing Motor Deficit
Description: No persistent new or increasing motor deficit
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 74 | 146
Participants | 72 | 144

8. Primary Outcome: Number of Subjects With no Reoperations or Epidural (Up to Day 1825)
Description: No reoperations, revisions, removals or supplemental fixation and no epidural injection at any lumbar level up to and including the Month 60 visit.
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 107 | 215
Participants | 71 | 149

9. Secondary Outcome: Number of Subjects With a Decrease in Zurich Claudication Questionnaire (ZCQ) Symptom Severity of at Least 0.5 Points
Description: ZCQ is a scale that measures physical function, symptom severity, and patient satisfaction for patients with spinal stenosis. Scores range from 1-5 with a higher score indicating worsening disability.
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 54 | 126
Participants | 40 | 100

10. Secondary Outcome: Number of Subjects With Decrease in Zurich Claudication Questionnaire (ZCQ) Physical Function of at Least 0.5 Points
Description: ZCQ is a scale that measures physical function, symptom severity, and patient satisfaction for patients with spinal stenosis.
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 54 | 126
Participants | 38 | 98

11. Secondary Outcome: Number of Subjects With Maintenance or Improvement in SF-12 Physical Function Component
Description: Assessment of the patient's Quality of Life as measured by SF-12. Scores range from 0 to 100, where a zero score indicates the lowest level of health. Success was defined as subjects who maintained or improved from their SF-12 score at baseline.
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 44 | 106
Participants | 34 | 93

12. Secondary Outcome: Number of Subjects With Maintenance or Improvement in SF-12 Mental Health Component
Description: as for outcome 11
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 44 | 106
Participants | 31 | 72

13. Secondary Outcome: Number of Subjects With a Decrease in VAS Back Pain of at Least 20mm
Description: Improvement of the Visual Analog Scale (VAS) for low back pain (on the 100 mm scale) compared to control group. On a scale of 0 to 100, 0 indicates no pain and 100 indicates worst pain imaginable.
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 53 | 124
Participants | 40 | 104

14. Secondary Outcome: Number of Subjects With Decrease VAS Worse Leg Pain of at Least 20mm
Description: Improvement of the Visual Analog Scale (VAS) for leg pain (on the 100 mm scale) compared to control group. On a scale of 0 to 100, 0 indicates no pain and 100 indicates worst pain imaginable.
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 53 | 124
Participants | 41 | 99

15. Secondary Outcome: Mean Oswestry Disability Index (ODI) Score
Description: Assessment of disability from low back pain as measured by ODI (Oswestry Disability Index) mean score in each treatment group at 5 years. On a scale of 0-100, a higher score represents increased disability.
Time Frame: 5 years
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 54 | 126
units on a scale | 26.1 (22.2) | 24.5 (20.5)

16. Secondary Outcome: Mean Visual Analog Scale Back Pain Score
Description: Assessment of Back Pain as measured by VAS mean score in each treatment group at 5 years. On a scale of 0-100mm, a higher score represents worse pain.
Time Frame: 5 years
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 54 | 124
mm | 29.0 (31.0) | 25.4 (27.6)

17. Secondary Outcome: Mean Visual Analog Scale Leg (Worse) Pain Score
Description: Assessment of Worse Leg Pain by VAS mean score in each treatment group at 5 years. On a scale of 0-100mm, a higher score represents worse pain.
Time Frame: 5 years
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 54 | 124
mm | 25.2 (31.2) | 22.8 (28.1)

18. Secondary Outcome: Mean Visual Analog Scale (VAS) Leg (Right) Pain Score
Description: Assessment of Right Leg Pain by VAS mean score in each treatment group at 5 years. On a scale of 0-100mm, a higher score represents worse pain.
Time Frame: 5 years
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 54 | 124
mm | 16.0 (24.5) | 14.9 (21.6)

19. Secondary Outcome: Mean Visual Analog Scale (VAS) Leg (Left) Pain Score
Description: Assessment of Left Leg Pain by VAS mean score in both treatment groups at 5 years. On a scale of 0-100mm, a higher score represents worse pain.
Time Frame: 5 years
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 54 | 124
mm | 17.0 (26.8) | 18.4 (27.0)

20. Secondary Outcome: Number of Subjects With a Decrease in VAS Right Leg Pain of at Least 20mm
Description: as for outcome 13
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 53 | 124
Participants | 36 | 90

21. Secondary Outcome: Number of Subjects With a Decrease in VAS Left Leg Pain of at Least 20mm
Description: as for outcome 13
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 53 | 122
Participants | 37 | 78

22. Secondary Outcome: Mean Zurich Claudication Questionnaire (ZCQ) Symptom Severity Score
Description: Assessment of symptom severity by ZCQ mean score in both treatment groups at 5 years. ZCQ is a scale that measures physical function, symptom severity, and patient satisfaction for patients with spinal stenosis. Scores range from 1-5 with a higher score indicating worsening disability.
Time Frame: 5 years
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 54 | 126
units on a scale | 2.17 (0.85) | 2.08 (0.84)

23. Secondary Outcome: Mean Zurich Claudication Questionnaire (ZCQ) Physical Function Score
Description: Assessment of physical function by ZCQ mean score in both groups at 5 years. ZCQ is a scale that measures physical function, symptom severity, and patient satisfaction for patients with spinal stenosis. Scores range from 1-5 with a higher score indicating worsening disability.
Time Frame: 5 years
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 54 | 126
units on a scale | 1.81 (0.79) | 1.67 (0.68)

24. Secondary Outcome: Mean Short Form-12 Physical Component Score
Description: Assessment of the patient's Quality of Life as measured by SF-12 mean score in both treatment groups at 5 years. Scores range from 0 to 100, where a zero score indicates the lowest level of health.
Time Frame: 5 years
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 47 | 118
units on a scale | 42.1 (12.6) | 42.1 (11.2)

25. Secondary Outcome: Mean Short Form-12 Mental Component Score
Description: as for outcome 24
Time Frame: 5 years
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 47 | 118
units on a scale | 54.8 (8.4) | 54.1 (9.7)

26. Secondary Outcome: Patient Survey: Satisfaction
Description: Subjects who responded "Very Satisfied" or "Somewhat Satisfied".
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 87 | 160
Participants | 72 | 151

27. Secondary Outcome: Patient Survey: Recommendation of Treatment
Description: Subjects who responded "Definitely Yes" or "Probably Yes"
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 87 | 160
Participants | 70 | 145

28. Secondary Outcome: Pain Management: Class II Narcotics Usage by Device Group
Description: Number of subjects using Class II narcotics
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 81 | 156
Participants | 17 | 32

29. Secondary Outcome: Pain Management: NSAIDs/ASA/Acetaminophen Usage by Device Group
Description: Number of subjects using NSAIDs/ASA/Acetaminophen
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 81 | 156
Participants | 24 | 55

30. Other Pre Specified Outcome: Mean Rotation (F to E) in Degrees - At Level(s) of Implant
Description: As determined by independent radiographic lab, this is the average measure of rotation (flexion to extension) at the index level(s) in both treatment groups at 5 years.
Time Frame: 5 years
Population: This analysis was performed at each level implanted. Since there were subjects with 2 levels implanted, the number of levels is greater than the number of patients.
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: Levels
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 81 | 149
Number analyzed (Levels) | 105 | 205
degrees | 0.98 (1.17) | 3.13 (3.43)

31. Other Pre Specified Outcome: Rotation (F to E) in Degrees - Below Level of Implant
Description: As determined by independent radiographic lab, this is the average measure of rotation (flexion to extension) at the level below the implant in both treatment groups at 5 years.
Time Frame: 5 years
Population: This analysis was performed at the level below the 1- or 2-level device construct in both groups.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 74 | 140
degrees | 5.62 (3.69) | 5.83 (4.17)

32. Other Pre Specified Outcome: Rotation (F to E) in Degrees - Above Level of Implant
Description: As determined by independent radiographic lab, this is the average measure of rotation (flexion to extension) at the level above the implant in both treatment groups at 5 years.
Time Frame: 5 years
Population: This analysis was performed at the level above the 1- or 2-level device construct in both groups.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 76 | 146
degrees | 3.59 (2.89) | 3.52 (3.16)

33. Other Pre Specified Outcome: Translation (mm) - At Level(s) of Implant
Description: As determined by independent radiographic lab, this is the average measure of translation at the index level(s) in both treatment groups at 5 years.
Time Frame: 5 years
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Levels
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 81 | 149
Number analyzed (Levels) | 103 | 204
mm | 0.23 (0.32) | 0.82 (0.84)

34. Other Pre Specified Outcome: Translation (mm) - Below Level of Implant
Description: As determined by independent radiographic lab, this is the average measure of translation at the level below the implant in both treatment groups at 5 years.
Time Frame: 5 years
Population: This analysis was performed at the level below the 1- or 2-level device construct in both groups.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 72 | 139
mm | 0.63 (0.57) | 0.64 (0.61)

35. Other Pre Specified Outcome: Translation (mm) - Above Level of Implant
Description: As determined by independent radiographic lab, this is the average measure of translation at the level above the implant in both treatment groups at 5 years.
Time Frame: 5 years
Population: This analysis was performed at the level above the 1- or 2-level device construct in both groups.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 74 | 145
mm | 0.69 (0.57) | 0.83 (0.80)

36. Other Pre Specified Outcome: Anterior Disc Height (mm) - At Level(s) of Implant
Description: As determined by independent radiographic lab, this is the average measure of anterior disc height at the index level(s) in both treatment groups at 5 years.
Time Frame: 5 years
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Levels
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 81 | 149
Number analyzed (Levels) | 108 | 205
mm | 8.13 (3.19) | 8.89 (3.68)

37. Other Pre Specified Outcome: Posterior Disc Height (mm) - At Level(s) of Implant
Description: As determined by independent radiographic lab, this is the average measure of posterior disc height at the index level(s) in both treatment groups at 5 years.
Time Frame: 5 years
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Levels
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 81 | 149
Number analyzed (Levels) | 108 | 205
mm | 4.56 (1.65) | 4.46 (1.89)

38. Other Pre Specified Outcome: Translation (F to E) in Percent (%) - At Level(s) of Implant
Description: As determined by independent radiographic lab, this is the percentage of translation at the index level(s) in both treatment groups at 5 years.
Time Frame: 5 years
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: percent
Units Other Than Participants: Levels
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 81 | 149
Number analyzed (Levels) | 105 | 205
percent | 0.69 (0.89) | 2.38 (2.43)

39. Other Pre Specified Outcome: Translation (F to E) in Percent (%) - Below Level of Implant
Description: As determined by independent radiographic lab, this is the percentage of translation at the level below the implant in both treatment groups at 5 years.
Time Frame: 5 years
Population: This analysis was performed at the level below the 1- or 2-level device construct in both groups.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 74 | 140
percent | 1.95 (1.95) | 1.97 (1.88)

40. Other Pre Specified Outcome: Translation (F to E) in Percent (%) - Above Level of Implant
Description: As determined by independent radiographic lab, this is the percentage of translation at the level above the implant in both treatment groups at 5 years.
Time Frame: 5 years
Population: This analysis was performed at the level above the 1- or 2-level device construct in both groups.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 76 | 146
percent | 2.07 (1.68) | 2.40 (2.31)

41. Other Pre Specified Outcome: Average Disc Height (mm) - At Level(s) of Implant
Description: As determined by independent radiographic lab, this is the average measure of disc height at the index level(s) in both treatment groups at 5 years.
Time Frame: 5 years
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Levels
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 81 | 149
Number analyzed (Levels) | 108 | 205
mm | 6.34 (2.09) | 6.67 (2.45)

42. Other Pre Specified Outcome: Change From Pre-Op Anterior Disc Height (mm) - At Level(s) of Implant
Description: As determined by independent radiographic lab, this is the average change from baseline for anterior disc height at the index level(s) in both treatment groups at 5 years.
Time Frame: 5 years
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Levels
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 81 | 149
Number analyzed (Levels) | 106 | 200
mm | -1.38 (1.58) | -1.32 (1.75)

43. Other Pre Specified Outcome: Change From Pre-Op Posterior Disc Height (mm) - At Level(s) of Implant
Description: As determined by independent radiographic lab, this is the average change from baseline for posterior disc height at the index level(s) in both treatment groups at 5 years.
Time Frame: 5 years
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Levels
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 81 | 149
Number analyzed (Levels) | 106 | 200
mm | -0.49 (1.19) | -0.72 (1.26)

44. Other Pre Specified Outcome: Change From Pre-Op Average Disc Height (mm) - At Level(s) of Implant
Description: As determined by independent radiographic lab, this is the average change from baseline for disc height at the index level(s) in both treatment groups at 5 years.
Time Frame: 5 years
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Levels
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 81 | 149
Number analyzed (Levels) | 106 | 200
mm | -0.93 (1.02) | -1.02 (1.24)

45. Other Pre Specified Outcome: Change From Post-Op Anterior Disc Height (mm) - At Level(s) of Implant
Description: As determined by independent radiographic lab, this is the average change from immediate post-op for anterior disc height at the index level(s) in both treatment groups at 5 years.
Time Frame: 5 years
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Levels
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 81 | 149
Number analyzed (Levels) | 108 | 205
mm | -1.82 (1.39) | -0.98 (2.06)

46. Other Pre Specified Outcome: Change From Post-Op Posterior Disc Height (mm) - At Level(s) of Implant
Description: As determined by independent radiographic lab, this is the average change from immediate post-op for posterior disc height at the index level(s) in both treatment groups at 5 years.
Time Frame: 5 years
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Levels
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 81 | 149
Number analyzed (Levels) | 108 | 205
mm | -0.85 (1.00) | -1.90 (1.65)

47. Other Pre Specified Outcome: Change From Post-Op Average Disc Height (mm) - At Level(s) of Implant
Description: As determined by independent radiographic lab, this is the average change from immediate post-op for disc height at the index level(s) in both treatment groups at 5 years.
Time Frame: 5 years
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Levels
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 81 | 149
Number analyzed (Levels) | 108 | 205
mm | -1.33 (0.97) | -1.44 (1.47)

48. Other Pre Specified Outcome: Disc Angle in Degrees - At Level(s) of Implant
Description: As determined by independent radiographic lab, this is the mean disc angle at the index level(s) in both treatment groups at 5 years.
Time Frame: 5 years
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: Levels
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 81 | 149
Number analyzed (Levels) | 111 | 205
degrees | 6.02 (4.64) | 7.28 (5.19)

49. Other Pre Specified Outcome: Change From Pre-Op Disc Angle in Degrees - At Level(s) of Implant
Description: As determined by independent radiographic lab, this is the mean change in disc angle from baseline at the index level(s) in both treatment groups at 5 years.
Time Frame: 5 years
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: Levels
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 81 | 149
Number analyzed (Levels) | 109 | 200
degrees | -1.41 (3.10) | -1.00 (2.91)

50. Other Pre Specified Outcome: Change From Post-Op Disc Angle in Degrees - At Level(s) of Implant
Description: As determined by independent radiographic lab, this is the mean change in disc angle from immediate post-op at the index level(s) in both treatment groups at 5 years.
Time Frame: 5 years
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: Levels
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 81 | 149
Number analyzed (Levels) | 111 | 205
degrees | -1.57 (2.25) | 1.56 (3.82)

51. Other Pre Specified Outcome: Change From Post-Op Spondylolisthesis (mm) - At Level(s) of Implant
Description: As determined by independent radiographic lab, this is the measure of spondylolisthesis at the index level(s) in both treatment groups at 5 years.
Time Frame: 5 years
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Levels
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 81 | 149
Number analyzed (Levels) | 108 | 205
mm | -1.08 (3.37) | -1.01 (3.78)

52. Other Pre Specified Outcome: Change From Post-Op Spondylolisthesis (%) - At Level(s) of Implant
Description: As determined by independent radiographic lab, this is the measure of the percentage of spondylolisthesis at the index level(s) in both treatment groups at 5 years.
Time Frame: 5 years
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: percent
Units Other Than Participants: Levels
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 81 | 149
Number analyzed (Levels) | 108 | 205
percent | -3.4 (9.9) | -3.2 (11.2)

53. Other Pre Specified Outcome: Change From Pre-Op Spondylolisthesis (mm) - At Level(s) of Implant
Description: As determined by independent radiographic lab, this is the mean change in measure of spondylolisthesis at the index level(s) in both treatment groups at 5 years.
Time Frame: 5 years
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Levels
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 81 | 149
Number analyzed (Levels) | 106 | 200
mm | -0.12 (2.28) | -0.56 (1.82)

54. Other Pre Specified Outcome: Change From Post-Op Spondylolisthesis (mm) - At Level(s) of Implant
Description: As determined by independent radiographic lab, this is the mean change in measure of spondylolisthesis from immediate post-op at the index level(s) in both treatment groups at 5 years.
Time Frame: 5 years
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Levels
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 81 | 149
Number analyzed (Levels) | 108 | 205
mm | -0.77 (1.92) | -0.44 (1.91)

55. Other Pre Specified Outcome: Foraminal Height (X-ray) (mm) - At Level(s) of Implant
Description: This is the mean foraminal height via x-ray at the index level(s) in both treatment groups at 5 years.
Time Frame: 5 years
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Levels
Arm/Group | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 149
Number analyzed (Levels) | 205
mm | 17.33 (2.75)

56. Other Pre Specified Outcome: Change From Pre-Op Foraminal Height (X-ray) (mm) - At Level(s) of Implant
Description: This is the mean change in foraminal height via x-ray from baseline at the index level(s) in both treatment groups at 5 years.
Time Frame: 5 years
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Levels
Arm/Group | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 149
Number analyzed (Levels) | 200
mm | -0.47 (1.29)

57. Other Pre Specified Outcome: Change From Post-Op Foraminal Height (X-ray) (mm) - At Level(s) of Implant
Description: This is the mean change in foraminal height via x-ray from immediate post-op at the index level(s) in both treatment groups at 5 years.
Time Frame: 5 years
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Levels
Arm/Group | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 149
Number analyzed (Levels) | 205
mm | -1.81 (1.74)

58. Other Pre Specified Outcome: Bony Bridging
Description: Bridging through the posterolateral gutters, between the facet joints, between transverse processes, and/or between facet joint and transverse process will all be considered acceptable forms of bridging bone.
Time Frame: 5 years
Population: as for outcome 30
Measure: Count of Units; unit: Levels
Units Other Than Participants: Levels
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 81 | 149
Number analyzed (Levels) | 111 | 209
Levels
  NA | 0 | 209
  No | 17 | 0
  Yes | 84 | 0
  Indeterminate | 10 | 0

59. Other Pre Specified Outcome: Heterotopic Ossification
Description: Assessment applicable to coflex arm only. The assessment applies to bony formations that occur in and around the implant.
Time Frame: 5 years
Population: as for outcome 30
Measure: Number; unit: participants
Units Other Than Participants: Levels
Arm/Group | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 149
Number analyzed (Levels) | 209
participants
  NA | 0
  None | 91
  Grade I | 0
  Grade II | 24
  Grade III | 73
  Bony Bridging | 3
  Indeterminate | 18

60. Other Pre Specified Outcome: Fusion Status
Description: The assessment is an analysis of three component factors: Bridging Bone, Angular Motion and Translational Motion.
Time Frame: 5 years
Population: as for outcome 30
Measure: Count of Units; unit: Levels
Units Other Than Participants: Levels
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 81 | 149
Number analyzed (Levels) | 111 | 209
Levels
  NA | 0 | 0
  Not fused | 19 | 196
  Fused | 78 | 3
  Indeterminate | 14 | 10

61. Other Pre Specified Outcome: Interface Remodeling - At Level(s) of Implant
Description: Per level; Assessment applicable to coflex arm only. This is an assessment of the bone-implant interface.
Time Frame: 5 years
Population: as for outcome 30
Measure: Count of Units; unit: Levels
Units Other Than Participants: Levels
Arm/Group | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 149
Number analyzed (Levels) | 209
Levels
  NA | 0
  None | 75
  Mild | 70
  Moderate | 16
  Severe | 20
  Indeterminate | 28

62. Other Pre Specified Outcome: Device Condition (Coflex Arm)
Description: Per level; Assessment only applicable to coflex group. Device Condition in the investigational subjects was graded as: Intact, Deformed, Fractured, Migrated, or Dislodged.
Time Frame: 5 years
Population: as for outcome 30
Measure: Count of Units; unit: Levels
Units Other Than Participants: Levels
Arm/Group | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 149
Number analyzed (Levels) | 209
Levels
  NA | 0
  Intact | 184
  Deformed | 0
  Fractured | 3
  Migrated | 11
  Dislodged | 0
  Indeterminate | 11

63. Other Pre Specified Outcome: Device Condition (Fusion Control)
Description: Per level; This assessment is applicable to the fusion arm only. Device Condition in the control subjects will be graded as: Intact, Loose Screws, or Failed Hardware.
Time Frame: 5 years
Population: as for outcome 30
Measure: Count of Units; unit: Levels
Units Other Than Participants: Levels
Arm/Group | Posterolateral Fusion w/Pedicle Screws
Number analyzed (Participants) | 81
Number analyzed (Levels) | 111
Levels
  NA | 0
  Intact | 90
  Failed Graft | 0
  Loose Screws | 10
  Fractured Hardware | 2
  Indeterminate | 9

64. Other Pre Specified Outcome: Device Mobility
Description: Per level; Assessment is applicable to coflex arm only. Device Mobility is an expected occurrence in some subjects and represents the amount of the of lift-off of the implant from the inferior spinous process.
Time Frame: 5 years
Population: as for outcome 30
Measure: Count of Units; unit: Levels
Units Other Than Participants: Levels
Arm/Group | Coflex Interlaminar Technolgy
Number analyzed (Participants) | 149
Number analyzed (Levels) | 209
Levels
  NA | 0
  < 5 mm | 181
  >= 5 mm | 15
  Indeterminate | 13

ADVERSE EVENTS:
Time Frame: 5 years
Description: In place of serious adverse event (SAE), this study used Severe AE (reported in SAE section as device related Severe AE):
  * is life threatening
  * results in permanent impairment of a body function or permanent damage to a body structure; or
  * necessitates medical or surgical intervention to preclude permanent impairment of a body function or permanent damage to a body structure
Arm/Group | Posterolateral Fusion w/Pedicle Screws | Coflex Interlaminar Technolgy
All-Cause Mortality (participants affected / at risk) | 0/107 | 0/215
Serious Adverse Events (participants affected / at risk) | 64/107 | 109/215
Other Adverse Events (participants affected / at risk) | 101/107 | 199/215
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Posterolateral Fusion w/Pedicle Screws (N=107) | Coflex Interlaminar Technolgy (N=215)
Component Loosening (Musculoskeletal and connective tissue disorders) | 5 | 3
Component Breakage (Musculoskeletal and connective tissue disorders) | 1 | 0
Tear > 5mm (Musculoskeletal and connective tissue disorders) | 1 | 0
Fracture (Musculoskeletal and connective tissue disorders) | 1 | 4
Hematoma Requiring Drainage (Musculoskeletal and connective tissue disorders) | 1 | 0
Infection (deep) (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain; new, increased frequency, or worsening (Musculoskeletal and connective tissue disorders) | 19 | 29
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 2 | 0
Wound problems (Musculoskeletal and connective tissue disorders) | 2 | 6
Other (Metabolism and nutrition disorders) | 11 | 10
Cancer/Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 5
Cardiovascular (Cardiac disorders) | 5 | 17
Eye, Ear, Nose and Throat (EENT) (Ear and labyrinth disorders) | 1 | 1
Endocrine/Metabolic (Endocrine disorders) | 2 | 4
Gastrointestinal (Gastrointestinal disorders) | 6 | 10
Genitourinary (General disorders) | 5 | 5
Hematological (Blood and lymphatic system disorders) | 0 | 1
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 16 | 32
Neurological (Nervous system disorders) | 4 | 5
Psychiatric/Substance Abuse (Psychiatric disorders) | 3 | 0
Respiratory (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Skin and Subcutaneous (Skin and subcutaneous tissue disorders) | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Posterolateral Fusion w/Pedicle Screws (N=107) | Coflex Interlaminar Technolgy (N=215)
Component Loosening (Musculoskeletal and connective tissue disorders) | 2 | 1
Component Migration (Musculoskeletal and connective tissue disorders) | 1 | 3
Component Breakage (Musculoskeletal and connective tissue disorders) | 1 | 3
Incidental Durotomy (<= 5mm) (Musculoskeletal and connective tissue disorders) | 0 | 1
Fracture (Musculoskeletal and connective tissue disorders) | 1 | 8
Nerve Injury (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain; new, increased frequency, or worsening (Musculoskeletal and connective tissue disorders) | 29 | 61
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Wound problems (Musculoskeletal and connective tissue disorders) | 9 | 24
Other (Musculoskeletal and connective tissue disorders) | 20 | 46
Cancer/Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 6
Cardiovascular (Cardiac disorders) | 11 | 15
Eye, Ear, Nose, Throat (EENT) (Ear and labyrinth disorders) | 4 | 8
Endocrine/Metabolic (Endocrine disorders) | 5 | 10
Gastrointestinal (Gastrointestinal disorders) | 11 | 11
Genitourinary (General disorders) | 8 | 11
Hematological (Blood and lymphatic system disorders) | 6 | 7
Immune (Immune system disorders) | 0 | 2
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 65 | 119
Neurological (Nervous system disorders) | 23 | 56
Psychiatric/Substance abuse (Psychiatric disorders) | 5 | 1
Respiratory (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Skin and Subcutaneous Tissue (Skin and subcutaneous tissue disorders) | 9 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No